CLINICAL TRIAL: NCT04817436
Title: Effects of Adapated Physical Activity Program on Kynurenin Metabolism During Refeeding in Anorexia Nervosa : APANOR Study
Acronym: APANOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/0383/HP
Record Dates: First submitted 2020-06-25; First posted 2021-03-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without adapted physical activity program (APA) (Active Comparator)
  Interventions: Other: physical activity program (APA)
- With adapted physical activity program (APA) (Experimental)
  Interventions: Other: physical activity program (APA)

INTERVENTIONS:
Other: physical activity program (APA) — adapted physical activity program (APA)

SUMMARY:
Physical hyperactivity is often associated to anorexia nervosa (AN). Data suggest common central pathways between hyperactivity and anorexia. Maintaining adapted physical activity (APA) during refeeding in AN is controversial. Many studies suggest beneficits of APA in AN on body composition (increase fat free mass and better distribution of fat mass), mood regulation, bone metabolism. We recently reported benefits of maintaining physical activity during refeeding in a mice model of anorexia (activity-based anorexia model). These benefits involved the tryptophan-kynurenin pathway. Thus, we aim in the APANOR study to assess effects of APA during refeeding in AN on kynurenin metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Patient > 18 years
3. Follow-up in the department of clinical Nutrition of Rouen
4. BMI ≥15,0 and <18,5 kg/m²
5. Diagnosis of anorexia nervosa according to DSM-V classification

Exclusion Criteria:

1. Physical activity contraindications : hemodynamic disorder, uncontrolled cardiovascular disease, intracranial hypertension
2. Patients with poor understanding of spoken or written French
3. Person deprived of their liberty by an administrative or judicial decision or person subject to a legal measure for the protection of adults
4. Person subject to a safeguard of justice, guardianship or curatorship.
5. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of adapated physical activity (APA) program on kynurenin metabolism | 3 months
  Variation of plasmatic kynurenin acid between V1 and V2 in patients undergoing APA during refeeding versus other patients (control group without APA)

SECONDARY OUTCOMES:
To evaluate the effects of adapated physical activity program on anthropometric data. | 3 months
  Anthropometric data
To evaluate the involving of gut microbiota composition and diversity | 3 months
  gut microbiota analyses
To evaluate the effects of adapated physical activity program on quality of life | 3 months
  Self-administered questionnaires assessing the quality of life
To evaluate the involving of auto-antibodies against neuropeptides involved in food intake regulation | 3 months
  Dosage of auto-antibodies against neuropeptides involved in food intake regulation using ELISA method (enzyme-linked immunosorbent assay)
To evaluate the effects of adapated physical activity program on Body composition (fat mass, fat free mass) | 3 months
  Mesaurement of fat and free mass

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Rouen, Rouen, France